CLINICAL TRIAL: NCT01108640
Title: Continuous Glucose Monitoring in Critically Ill Surgical Patients
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 0912006043
Record Dates: First submitted 2010-04-07; First posted 2010-04-22 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Hyperglycemia
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Elective surgical patients
- Massive resuscitation patients
- surgical patients on pressors

SUMMARY:
The specific aim of this study is to identify the degree of correlation between real time subcutaneous glucose monitoring and intermittent glucose monitoring using capillary glucose samples, arterial blood samples and venous blood samples in critically ill surgical patients. A secondary aim will be to determine the accuracy of real time glucose monitoring.

DETAILED DESCRIPTION:
Patients:

This study will be conducted in the surgical intensive care unit (SICU) at Yale New Haven Hospital in a prospective observational fashion. As this is a pilot study to determine the accuracy of CGM in our patient population we have based our enrollment projection to complete the study within an approximately 8 month time frame. We will identify three groups of 15 patients who are candidates for enrollment. The primary outcome is the degree of correlation between the continuous glucose monitor and capillary or arterial blood samples.

The first group will be patients who present to the SICU and are hemodynamically unstable. Hemodynamic instability will be defined as systolic blood pressure less than 90 mmHg or the requirement of continuous infusion of vasopressors to maintain the systolic blood pressure over 90 mmHg. The second group of patients will be a similar group that is expected to require massive fluid or blood resuscitation (>6L crystalloid or >6 units of blood) to maintain systolic blood pressure over 90 mmHg. This second group of patients will consist mainly of trauma patients. These patients or their closest available relative will be approached for consent to participate in the trial. For patients enrolled through a surrogate who regain their decision making capacity they will be informed of their participation in the study by one of the investigators.

The third group will be patients undergoing elective surgical procedures that will likely require a post-operative admission to the SICU. This group will include patients undergoing open abdominal aortic aneurysm repair, esophagectomy, or other major abdominal or thoracic operation that will likely require a SICU stay of more than 24 hours. At least half of this group will consist of diabetic patients. These patients will be selected by one of the investigators based on their likelihood of requiring more than 24 hours of SICU care. Based on the experience of the investigators we believe we will be able to accurately predict which patients will require an ICU stay of at least 24 hours. Most commonly these patients will have significant co-morbid medical conditions including coronary artery disease, hypertension, hypercholesterolemia, obesity, etc. An attempt will be made to contact these patients pre-operatively by telephone within 1 week of their planned surgery at which time details of the research will be explained. Their willingness to participate will be ascertained and they will be formally enrolled and sign consent on the morning of surgery if possible. On some occasions patients will require ICU stays post-operatively that were not predicted pre-operatively. These patients and any patients that were not identified pre-operatively by the research team will be enrolled post-operatively often through their surrogate similar to the other study groups. Similarly if patient are enrolled pre-operatively and subsequently do not require SICU admission they will not undergo any of the study procedures and not be counted towards the total enrollment.

Study Procedures:

Upon arrival in the surgical ICU a subcutaneous glucose sensor (Guardian RT® CGMS) will be placed by one of the investigators after informed consent has been obtained. Insertion will be in the lower lateral abdomen using the insertion device provided with the Guardian RT® system. For patients for whom lower abdominal insertion is impossible, e.g. those with open abdomens, a site will be chosen in the proximal thigh or proximal arm based on the estimated thickness of the subcutaneous fat. The sensor transmits a signal wirelessly to a receiver/monitor. This receiver/monitor will be maintained in the patient's room. The meter will be calibrated based on an arterial or capillary blood glucose obtained within one hour of sensor insertion per pre-existing SICU routine care. The meter will then be recalibrated every 12 hours based on blood glucose measurements obtained per existing SICU routine. The existing protocol in the SICU is measurement of a blood glucose every hour while on an insulin infusion until stable then every 2 hours thereafter. For patients requiring only sub-cutaneous insulin blood glucose is measured at a minimum of every 4 hours. If necessary the sensor will be replaced a maximum of three times within 12 hours before placement will be considered a failure. Capillary or arterial blood glucose will be measured every hour if the patient is requiring a fluctuating insulin infusion. If the patient is on a stable insulin infusion blood glucose samples will be obtained every 2 hours. If the patient is not on an insulin infusion glucose levels will be obtained at least every 4 hours per pre-existing SICU protocols. All arterial or capillary glucose levels will be entered into the Guardian RT® system. Blood glucose measurements will be per the SICU routine. All SICU staff, physicians and study personnel will be blinded to the CGMS readings. Sensors will be changed after 72 hours and when the system identifies a problem with the sensor that can not be corrected through standard system diagnostics per manufacturer recommendations. Total attempts at sensor placement will be limited to a maximum of 4 over the course of each subject's participation in the study. Sensors will be removed when the patient is transferred from the SICU, if the patient expires, or if the patient's care is transitioned to comfort measures only. At the end of the second sensor life-time (144 hours) the sensor will be removed and data collection will be terminated.

In addition to the glucose data, administration of all insulin and other medications likely to affect blood glucose levels or perfusion status will be recorded as will all infusions containing dextrose, including parenteral nutrition and all enteral feeding. All other clinical events such as return trips to the operating room, or development of a new infection, or new organ failure, will be recorded by the investigative team. Additional data collected will include age, gender, race, prior medical history, reason for SICU admission, medications during the study and prior, complications, days on mechanical ventilation, length of stay, daily vital signs, including weight and any vital sign abnormalities, body mass index, liver failure, renal failure and use of renal replacement therapy. If a patient develops a skin reaction to the device or the adhesive maintaining the device, it will be removed and a new site will be employed if possible with tape replacing the standard transparent dressing.

Data analyses:

Data from each sensor will be downloaded and blood glucose values obtained using proprietary software from Medtronic. Because the CGMS system records glucose readings every 5 minutes capillary or arterial glucose samples obtained will be compared with the closest CGMS reading within 2.5 minutes of the time the sample was obtained. This will generate a set of paired glucose levels for analysis. If the sample falls immediately between 2 readings the later of the CGMS readings will be used to minimize the effect of the lag time for interstitial glucose.

Several methods will be used to assess accuracy of the CGMS. The International Organization for Standardization (ISO) has put forth requirements for blood glucose monitoring systems. For reference values ≤75mg/dl sensor values should be within ±15mg/dl, and for reference values >75mg/dl sensor values should be within ±20%. We will initially determine the percentage of glucose pairs that meet these criteria. To determine the degree of agreement between sensor and reference the mean difference (MD, average of sensor values - reference values), mean relative difference (MRD, MD divided by the reference value multiplied by 100) will be calculated. The MD and MRD allow determination of a general under or overestimation by the sensor. The mean absolute difference (MAD, mean of the absolute value of: sensor value - reference value) will be calculated. The mean and median absolute relative difference (ARD, mean and median of the absolute value of: (sensor value - reference value) *100 / reference value) will also be calculated. These absolute differences provide insight into the overall accuracy of each individual meter reading. In the previous study in the medical intensive care unit 22 patients resulted in 546 glucose pairs for analysis. The calculated MAD was 19.7 with a standard deviation of 18.3. This resulted in a 95% confidence interval of [18.2-21.2]. In our study if we use a relatively conservative estimate of 45 patients studied for 1 day (24 hours) each with blood glucose measurements every 2 hours this results in 540 meter-sensor glucose pairs. Based on these data our study will result in a similarly narrow confidence interval for the MAD.

Bland-Altman plots will be constructed. These are plots of the difference between the values of each glucose pair (y-axis) versus the average of the two members of the pair (x-axis). These plots are helpful to identify particular areas of inaccuracy in the range of glucose reading e.g. at very high or very low glucose levels. The accuracy of the reference reading must be considered when analyzing these plots.

Clarke error grids have become one of the most accepted methods of analyzing continuous glucose data. These grids are plots of the CGMS reading versus the reference value. Areas on the grid are constructed based on the clinical effects of each paired blood glucose. The paired glucose readings are thereby classified as in good agreement or erroneous with varying levels of clinical consequence. In order to identify inaccuracy based on the time delay of the CGMS we will randomly select one or two multiple hour time periods from each patient. We will compare plots of the CGMS readings with time shifted plots of the capillary or arterial blood glucose readings and attempt to obtain matches to identify the effect of the time delay. We will also analyze the effect of fluid loading and interstitial edema on the accuracy of the meters as well as the time delay.

We will define significant interstitial edema as an increase in body mass by 15% or more above admission body weight.

It is anticipated that we will be able to enroll 2 patients per month in each group generating study enrollment duration of at least 8 months. Enrollment in this fashion will require approximately 5 monitors and 75 sensors.

ELIGIBILITY:
Inclusion Criteria:

* Septic surgical patients,
* Surgical patients undergoing massive resuscitation,
* Elective surgical patients.

Exclusion Criteria:

* Pregnancy,
* No safe location to place a sensor (skin disorder in areas of potential placement, minimal subcutaneous tissue),
* Patient/surrogate declines to participate,
* Patients speaking a language other than English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to a surgical intensive care unit and falling into one of the three groups
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Concordance of continuous glucose monitor with standard capillary and arterial blood glucose | 9 months
  Data from each sensor will be downloaded and blood glucose values obtained using proprietary software from Medtronic. Because the CGMS system records glucose readings every 5 minutes, capillary or arterial glucose samples obtained will be compared with the closest CGMS reading within 2.5 minutes of the time the sample was obtained. This will generate a set of paired glucose levels for analysis.

SECONDARY OUTCOMES:
Safety of the sensor in terms of infection or bleeding at the insertion site | 9 months
  The monitor insertion site will be observed by the bedside nurse for infectious or bleeding complications

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Schuster, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Result] Schuster KM, Barre K, Inzucchi SE, Udelsman R, Davis KA. Continuous glucose monitoring in the surgical intensive care unit: concordance with capillary glucose. J Trauma Acute Care Surg. 2014 Mar;76(3):798-803. doi: 10.1097/TA.0000000000000127. PMID 24553551